CLINICAL TRIAL: NCT00084188
Title: HIV/STD Safer Sex Skills Groups for Women in Drug Treatment Programs
Brief Title: HIV/STD Safer Sex Skills Groups for Women in Drug Treatment Programs - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Susan Tross, Ph.D., New York State Psychiatric Institute
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTN-0019-1
Record Dates: First submitted 2004-06-08; First posted 2004-06-09 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Behavior Therapy
Keywords: behavioral intervention
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to look at a program for women in drug abuse treatment designed to reduce Human Immunodeficiency Virus/Sexually Transmitted Disease (HIV/STD) risk behaviors and reduce unprotected sexual risk behavior.

DETAILED DESCRIPTION:
The proposed trial is intended to test the effectiveness of a proven, manual driven, five-session safer sexual skills building group (SSB) intervention (Schilling et al., 1991; El Bassel and Schilling, 1992) for female patients in MMTP or in drug-free outpatient treatment. The effects of SSB will be compared to a standard group HIV education session (HE).

This study uses a 2-group, randomized, parallel-group design to compare a five-session safer sexual skills building group to a single 60-min HIV education session (control condition). The control condition is designed to standardize and simulate the usual care at community clinics.

ELIGIBILITY:
Adult females (18 years of age or older) in drug abuse treatment at participating Community Treatment Programs are invited to participate.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541
Dates: Start 2004-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
AIDS risk behavior

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tross, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (12):
- United States (12):
  - Baart Cdp, Los Angeles, California
  - Hartford Dispensary, New Britain, Connecticut
  - Staten Island University Hospital, Staten Island, New York
  - Addiction Drug Services, Greensboro, North Carolina
  - South Light - Life Plus, Raleigh, North Carolina
  - South Light - Wakeview, Raleigh, North Carolina
  - Comprehensive Addiction Services System, Toledo, Ohio
  - The Consortium, Philadelphia, Pennsylvania
  - Thomas Jefferson Intensive Sub. Abuse TP, Philadelphia, Pennsylvania
  - LRADAC-Lexington-Richmond Alcohol & Drug Council, Columbia, South Carolina
  - Evergreen Treatment Services, Seattle, Washington
  - Prestera Center for Mental Health Svcs., Huntington, West Virginia

REFERENCES:
- [Derived] Campbell AN, Tross S, Hu MC, Pavlicova M, Kenney J, Nunes EV. Female condom skill and attitude: results from a NIDA Clinical Trials Network gender-specific HIV risk reduction study. AIDS Educ Prev. 2011 Aug;23(4):329-40. doi: 10.1521/aeap.2011.23.4.329. PMID 21861607
- [Derived] Tross S, Campbell AN, Cohen LR, Calsyn D, Pavlicova M, Miele GM, Hu MC, Haynes L, Nugent N, Gan W, Hatch-Maillette M, Mandler R, McLaughlin P, El-Bassel N, Crits-Christoph P, Nunes EV. Effectiveness of HIV/STD sexual risk reduction groups for women in substance abuse treatment programs: results of NIDA Clinical Trials Network Trial. J Acquir Immune Defic Syndr. 2008 Aug 15;48(5):581-9. doi: 10.1097/QAI.0b013e31817efb6e. PMID 18645513